CLINICAL TRIAL: NCT04066699
Title: Intraoperative, Percutaneous Localization of Peripheral Pulmonary Nodules for Resection: a Prospective, Open-Label, Multi-Center Registry Study of Thoracic Surgery Outcomes.
Brief Title: Percutaneous Localization: Open-label Registry of Thoracic Surgery
Acronym: PLOTS
Status: Completed | Type: Observational
Sponsor: Veran Medical Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: VMT-01-003
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Lung Lesion(s) Requiring Evaluation; Pulmonary Metastasis; Pulmonary Nodule, Solitary; Peripheral Lung Lesions
Keywords: Surgical Lung Resection; Percutaneous Localization; Electromagnetic Navigation; Transthoracic Localization; Peripheral Pulmonary Nodule(s)
MeSH Terms: conditions — Solitary Pulmonary Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Localization: Electromagnetic navigation (EMN) guided percutaneous localization of suspicious lung lesion(s).
  Interventions: Procedure: Percutaneous localization of suspicious lung lesion(s) using electromagnetic navigation and tools.

INTERVENTIONS:
Procedure: Percutaneous localization of suspicious lung lesion(s) using electromagnetic navigation and tools. — Transthoracic localization of suspicious lung lesion(s) in preparation for subsequent resection.
  Other Names: SPiN Thoracic Navigation System™; Veran System

SUMMARY:
The objectives of this study are to evaluate intraoperative percutaneous lung lesion marking assisted by electromagnetic guided percutaneous navigation and related tools.

DETAILED DESCRIPTION:
The Intraoperative, Percutaneous Localization of Peripheral Pulmonary Nodules for Resection: a Prospective, Open-Label, Multi-Center Registry Study of Thoracic Surgery Outcomes (PLOTS) registry is aimed at developing a high quality set of data regarding intraoperative percutaneous localization of peripheral pulmonary nodules (PPNs), and then identifying and promulgating efficient, evidence-based best practices for this technique. The resection procedure itself is standard of care and follows the investigator's standard protocol.

Successful localization of PPNs is a challenge involving multiple factors, beginning with the subjects' health, lung function and also factors specific to the nodule including location within the lung, size, distance from the lung surface, whether solid or ground glass and proximity to a fissure. Hard to see or palpate nodules are currently localized with dye and/or hook wires or fiducials, either endoscopically or percutaneously. Successful, large, prospective studies have not been reported using modern electro-magnetic navigation (EMN)-guided percutaneous intraoperative localization, and different techniques (dye vs. fiducial vs. hook wire etc.) have not been broadly evaluated. It is for these reasons that the different localization techniques used with EMN-guided percutaneous localization will be collected for patients having a suspicious nodule and who undergo percutaneous intra-operative localization and immediate resection.

This registry aims to record the localization techniques used by thoracic surgeons and IP/surgical teams to identify PPNs using the SPiN Thoracic Navigation System™ in the hands of trained physicians. The objectives of this study will be to accomplish the primary and secondary objectives listed below, and to observe localization in a real world context of pulmonary resection.

ELIGIBILITY:
Inclusion Criteria:

* Subject's physician and/or thoracic surgeon have deemed/has deemed that the surgical removal of the PPN is appropriate.
* A clinical decision has been made to use the SPiN Thoracic Navigation System™.
* Subject is at least 18 years of age at time of study entry.
* Subject is able to read, understand, and voluntarily sign the IRB-approved informed consent document prior to the performance of any study-specific procedures. IRB- approved translation may be used if indicated. Reasonable accommodation of visually impaired subjects will be allowed.
* Subject is able to tolerate general anesthesia.
* Subject has a target nodule between 0.4 cm and 3.2 cm in greatest dimension;
* The target nodule is in a location that is accessible for percutaneous localization in the judgement of the surgeon.

Exclusion Criteria:

* Subjects with any other concomitant treatment or medical condition that, in the opinion of the clinician, would render peripheral nodule resection more hazardous than beneficial.
* Subject is pregnant.
* Pulmonary nodule is greater than 3.2 cm.
* Subjects with significant coagulopathy having INR > 2.0 or PTT > 2x normal.
* Subject is unable to tolerate general anesthesia.
* Obese subject, impacting percutaneous access (BMI > 50).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target subject population includes adult subjects (18 years - 85 years), with small, suspicious lung lesions. Patients with small, indeterminate PPNs that, in the judgment of the thoracic surgeon, based on surgical risk and risk of malignancy, warrant lung resection via a percutaneous localization approach. Data will be collected from study subjects having a PPN between 0.4 cm and 3.2 cm in greatest dimension, that are accessible to percutaneous localization, who consent to and undergo intraoperative dye/wire localization procedure followed by surgical lung resection.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Rate of successful percutaneous localization and removal of PPN. | Duration of procedure.
  Successful percutaneous localization of PPN defined as the percentage of subjects in whom the nodule is successfully localized and removed in the first resected specimen.
Safety of the localization procedure. | Duration of procedure.
  Safety data, including instances of adverse events and device deficiencies, will be collected.

SECONDARY OUTCOMES:
Localization method and technique. | Duration of procedure.
  Details regarding the localization technique will be collected, including the materials used. If dye (methylene blue, ICG etc.) is used the volume will be collected. Other materials include microcoils, hook wires, etc..
Intraoperative percutaneous localization time and duration of total surgical procedure. | Duration of procedure.
  The time of the localization procedure will be recorded. The length of the entire surgical procedure will also be recorded.
Nodule characteristics, including location in the lobe, distance from pleura, distance from surface of skin to target, morphological appearance, solid vs. ground glass etc. | Duration of procedure.
  Details regarding nodule characteristics - solid, semisolid, groundglass; location in relation to anatomical markers and position; size; presence of spiculation - will be collected.
Weight of excised tissue and margin. | Duration of procedure.
  The weight (in grams) of excised tissue will be recorded, as well as the measurement of the included margin.
Type of surgical resection performed and the resection technique used. | Duration of procedure.
  The surgical resection may include segmentectomy or wedge using the VATS, RATS, or thoracotomy techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Faiz Bhora, MD, Principal Investigator — Hackensack Meridian Health Network & School of Medicine
Locations (5):
- United States (5):
  - Kaiser Permanente, Lone Tree, Colorado
  - Northern Light Eastern Maine Medical Center, Bangor, Maine
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Houston Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Semaan RW, Lerner AD, Lee HJ, Feller-Kopman D, Yarmus LB. Electromagnetic Guidance for the Diagnosis of Pulmonary Nodules: Don't Put the Nail in the Coffin. Am J Respir Crit Care Med. 2016 Jul 1;194(1):121. doi: 10.1164/rccm.201602-0243LE. No abstract available. PMID 27367891
- [Background] Mallow C, Lee H, Oberg C, Thiboutot J, Akulian J, Burks AC, Luna B, Benzaquen S, Batra H, Cardenas-Garcia J, Toth J, Heidecker J, Belanger A, McClune J, Osman U, Lakshminarayanan V, Pastis N, Silvestri G, Chen A, Yarmus L. Safety and diagnostic performance of pulmonologists performing electromagnetic guided percutaneous lung biopsy (SPiNperc). Respirology. 2019 May;24(5):453-458. doi: 10.1111/resp.13471. Epub 2019 Jan 24. PMID 30675961
- [Background] Thiboutot J, Lee HJ, Silvestri GA, Chen A, Wahidi MM, Gilbert CR, Pastis NJ, Los J, Barriere AM, Mallow C, Salwen B, Dinga MJ, Flenaugh EL, Akulian JA, Semaan R, Yarmus LB. Study Design and Rationale: A Multicenter, Prospective Trial of Electromagnetic Bronchoscopic and Electromagnetic Transthoracic Navigational Approaches for the Biopsy of Peripheral Pulmonary Nodules (ALL IN ONE Trial). Contemp Clin Trials. 2018 Aug;71:88-95. doi: 10.1016/j.cct.2018.06.007. Epub 2018 Jun 7. PMID 29885373

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT04066699/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT04066699/ICF_001.pdf